CLINICAL TRIAL: NCT05410782
Title: A Three Month Course of Power Prenatal Supplements to Improve Sperm Quality in Male-factor Infertility Patients
Brief Title: Power Prenatal Supplements for Sperm Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Bird and Be Co Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Power Prenatal for Sperm
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-08

CONDITIONS: Spermatogenesis and Semen Disorders; Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Sperm Count; Prenatal Care

STUDY DESIGN:
Intervention Model Description: Patients with male factor infertility, who have a document abnormal semen analysis (at least 1 of 3 abnormal parameters - concentration, progressive motility or morphology) will be recruited to take a 3 month course of supplements (Power Prenatal for Sperm), and a repeat semen analysis will be performed after the intervention to compare results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Power Prenatal for Sperm (Experimental): This is a single arm study. Participants will take supplements for 3 months. The supplements is Power Prenatal for Sperm (active ingredients - https://birdandbe.com/the-power-prenatal-for-sperm)
  Interventions: Dietary Supplement: Power Prenatal for Sperm

INTERVENTIONS:
Dietary Supplement: Power Prenatal for Sperm — A prenatal vitamin complex that includes numerous ingredients aim at improving sperm quality (ingredients: https://birdandbe.com/the-power-prenatal-for-sperm)
  Other Names: Prenatal Vitamins

SUMMARY:
Male factor infertility is a leading cause of primary and secondary infertility. Poor sperm quality is defined as having an abnormal semen analysis [WHO 2020 - https://www.who.int/publications/i/item/9789240030787]. The effects of supplements (vitamins, minerals, and anti-oxidants) on improving sperm quality are still debated (https://pubmed.ncbi.nlm.nih.gov/30462179). Taking additional supplements to improve sperm quality represent a modifiable risk-factor that would be an easy intervention for patients struggling with male factor infertility. The life cycle of sperm production is estimated at 3 months, so any intervention would require a 3 month course to see its full effect.

The investigators hypothesize that a 90 day course of the "Power Prenatal for Sperm", a male fertility supplement by Bird&Be (https://birdandbe.com/the-power-prenatal-for-sperm) will improve sperm quality based on semen analysis results prior to, and after taking the supplements.

DETAILED DESCRIPTION:
Male patients presenting to Conceive Health (https://conceivehealth.com/) or Reproductive Care Centre for infertility care will be potential candidates for this study. Male patients that have had a recent abnormal semen analysis conforming at least 1 of 3 parameters (low concentration: < 15 Million / mL; low progressive motility < 30%, and low morphology with strict criteria < 4%) will be eligible to participate.

Patients will be approached by a study coordinator to participate in the study. The study coordinator will ensure all inclusion and exclusion criteria is met, consents forms are signed, and a 90 day course of the "Power Prenatal for Sperm" is dispensed

Study participants will be instructed to repeat a semen analysis (at the same lab) after their 90 day course of the "Power Prenatal for Sperm". The differences between the semen analysis parameters will be compared

The primary outcome was chosen as processive motility, as this parameter is mostly likely to be positively impacted by the Power Prenatal for Sperm.

An abnormal progressive motility is defined as <5th percentile (32%) of the semen analysis of the fertile male population. The standard deviation for this population is 13.5%. The estimated effect size is 37.5%, from 32% to 44%, an increase of 12%. The alpha (type 1 error) significant level was set at 5% and the power level was set at 80%. The required sample size was 40 patients. Given that this study requires a 3 month intervention prior to a follow up semen analysis for comparison, the investigators estimated a 20% drop-out rate, so the total requirement was set at 50 patients.

Table A1.2 (https://www.who.int/docs/default-source/reproductive-health/srhr-documents/infertility/examination-and-processing-of-human-semen-5ed-eng.pdf)

Statistical analyses will be performed using standard expected methods. All data will be presented as mean ± Standard Deviation (SD). Statistical significance between semen analysis data will be determined by using the Shapiro-Wilk test of normality for predictions and paired samples t-test.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-45 years old
* Experiencing infertility
* A recent semen analysis confirming low count, motility or morphology (at least 1 of 3) - within last 3 months

  1. Low concentration: < 15 Million / mL
  2. Low Motility: Progessive Motility < 30%
  3. Morphology: Strict criteria: Normal forms < 4% Reference: WHO 2020 6th edition: https://www.who.int/publications/i/item/9789240030787

Exclusion Criteria:

* No diagnosed varicocele
* Younger than 18 years old
* Older than 45 years old
* Currently taking any form of antioxidant supplements(in last 3 months) besides a general multivitamin

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sperm Progressive Motility (Semen Analysis); as percentage (%) | A repeat semen analysis will be performed 3 months after Power Prenatal for Sperm intervention
  Semen analysis

SECONDARY OUTCOMES:
Sperm Concentration (Semen Analysis); as millions / mL | A repeat semen analysis will be performed 3 months after Power Prenatal for Sperm intervention
  Semen analysis
Sperm Morphology (Semen Analysis); as percentage (%) | A repeat semen analysis will be performed 3 months after Power Prenatal for Sperm intervention
  Semen Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nayot, BSc, MSc, MD, Principal Investigator — The Bird and Be Co
Locations (1):
- Reproductive Care Centre, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No